CLINICAL TRIAL: NCT00758121
Title: CORRELATE-HF: Correlation Of Respiratory Rate Level And Trend Evaluation in Heart Failure Patients
Brief Title: Correlation Of Respiratory Rate Level And Trend Evaluation in Heart Failure Patients
Acronym: CORRELATE-HF
Status: Terminated | Type: Observational
Why Stopped: Inappropriate therapy associated with certain right ventricular (RV) lead complications may occur more frequently if the Respiratory Sensor is programmed On
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Steve McQuillan / Director, Clinical Affairs, Boston Scientific CRM
Other Study IDs: CR-CA-091008-H
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Last update posted 2009-11-06 (Estimated); Status verified 2009-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Heart failure patients with an implanted CRT-D
  Interventions: Device: Cardiac Resynchronization Therapy Defibrillator

INTERVENTIONS:
Device: Cardiac Resynchronization Therapy Defibrillator — CRT-D observational study

SUMMARY:
The objective of the study is to determine if there is any relationship between respiratory rate and Heart Failure events.

DETAILED DESCRIPTION:
The purpose of the CORRELATE-HF study is to collect RRT data in heart failure patients to gain a better understanding of how respiratory rate changes in relation to all cause clinical events as well as other diagnostic features, including but not limited to, activity level, heart rate, and lead impedance.

ELIGIBILITY:
Inclusion Criteria:

* Implanted COGNIS device or future commercially available Boston Scientific CRT-D, that contains the Sensor Trend for Respiratory Rate, with a right ventricular lead and left ventricular lead actively implanted
* Respiratory Sensor programmed "On"
* Classified as having NYHA Class III heart failure documented, in the past 12 months
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Willing and capable of providing informed consent, participating in all testing associated with this clinical investigation at an approved clinical investigational center and at the intervals defined by this protocol

Exclusion Criteria:

* Inability or refusal to sign the patient Informed Consent
* Inability or refusal to comply with the follow-up schedule
* Patients that have received routinely scheduled intravenous inotropic therapy as part of their drug regimen within the past 90 days
* Patients prescribed to positive airway pressure therapy
* A life expectancy of less than 180 days, per physician discretion
* Enrolled in any concurrent study without prior written approval from Boston Scientific CRM
* Women who are pregnant or plan to become pregnant in the next twelve months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with an implanted CRT-D.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jaski, MD, Principal Investigator — San Diego Cardiac Center; Pedro Brugada, MD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- San Diego Cardiac Center, San Diego, California, United States
- UZ Brussel, Brussels, Belgium